CLINICAL TRIAL: NCT03467178
Title: Randomized Phase II Study on Decitabine Plus Carboplatin Versus Physician's Choice Chemotherapy in Recurrent, Platinum-resistant Ovarian Cancer.
Brief Title: Study on Decitabine Plus Carboplatin Versus Physician's Choice Chemotherapy in Recurrent, Platinum-resistant Ovarian Cancer.
Acronym: MITO29
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT 189-17
Record Dates: First submitted 2018-02-16; First posted 2018-03-15 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Recurrent, Platinum-resistant Ovarian Cancer
MeSH Terms: conditions — Recurrence | interventions — Decitabine; Carboplatin; liposomal doxorubicin; Gemcitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decitabine plus Carboplatin (Experimental): Carboplatin AUC 5 d 8 q 28 plus Decitabine 10 mg/mq iv d1-5 q 28
  Interventions: Drug: Decitabine; Drug: Carboplatin
- Standard Treatment (Other): Pegylated Liposomal Doxorubicin 40 mg/mq q 28 or Gemcitabine 1000 mg/mq dd 1, 8, 15 q 28 or Weekly Paclitaxel 80 mg/ m2 dd 1, 8, 15 q 28
  Interventions: Drug: Pegylated Liposomal Doxorubicin; Drug: Gemcitabine; Drug: Paclitaxel

INTERVENTIONS:
Drug: Decitabine — Nucleic Acid Synthesis Inhibitor
  Arms: Decitabine plus Carboplatin
Drug: Carboplatin — Chemotherapy medication
  Arms: Decitabine plus Carboplatin
Drug: Pegylated Liposomal Doxorubicin — Chemotherapy medication
  Arms: Standard Treatment
Drug: Gemcitabine — Chemotherapy medication
  Arms: Standard Treatment
Drug: Paclitaxel — Chemotherapy medication
  Arms: Standard Treatment

SUMMARY:
Multicenter Phase II study on Decitabine-Carboplatin combination in platinum resistant ovarian cancer patients.

Patients will receive study treatment until disease progression is documented, extraordinary medical circumstances occur, intolerable toxicities occur, or the patient withdraws consent.

DETAILED DESCRIPTION:
This is an open-label, prospective, multicenter, randomized Phase II, clinical trial evaluating the efficacy and safety of Decitabine-Carboplatin combination in recurrent, platinum resistant ovarian cancer patients in comparison to physician' choice chemotherapy:

Arm A: Carboplatin AUC (Area Under Curve) 5 d 8 q 28 Plus Decitabine 10 mg/mq iv d1-5 q 28

Arm B: Pegylated Liposomal Doxorubicin 40 mg/mq q 28 or Gemcitabine 1000 mg/mq dd 1, 8, 15 q 28 or Weekly Paclitaxel 80 mg/mq gg 1, 8, 15 q 28

Patients will be randomly assigned in a 1:1 ratio to treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Cytologic / histologic diagnosis of stage 1°C-4° epithelial , fallopian tube and primary peritoneal cancer (carcinosarcomas are included)
* Patient who received 1-2 prior lines of treatments
* Patient relapsed within 6 months after platinum containing regimen
* Disease measurable or evaluable by RECIST version 1.1 or Ca 125 GCIG criteria (Gynaecologic Cancer Intergroup).
* No residual peripheral neurotoxicity > Grade 1 from previous chemotherapy treatment
* Performance Status (PS) 0-1
* Age 18 years.
* Life expectancy of at least 3 months
* Written informed consent prior to performance of study specific procedures or assessments
* Ability and willingness to comply with treatment and follow up assessments and procedures
* Adequate organ functions:

  1. Hematopoietic: Leukocytes > 2,500/mm3; Absolute neutrophil count >1,500/mm3; Platelets count >100,000/mm3; Hemoglobin >9 g/dL
  2. Hepatic: AST (aspartate transaminase ) and ALT (alanine transaminase) <3 times upper limit of normal (ULN)*; Alkaline phosphatase <3 times ULN*; Bilirubin <1.5 times ULN

     *: <5 times ULN if liver metastases are present
  3. Renal: Creatinine clearance >45 mL/min
* No other invasive malignancy within the past 3 years except non-melanoma skin cancer and in situ cervical cancer
* Absence of any psychological, familial, sociological or geographical conditions potentially hampering compliance with the study protocol and follow-up schedule.

Exclusion Criteria:

* Pregnant (potentially fertile patients must use contraceptive measures to avoid pregnancy during and for at least 3 months after study participation and must have a negative serum pregnancy test at baseline).
* Patients should not be breast-feeding during treatment and for 2 months following the end of treatment.
* Serious heart disease, including heart failure, atrio-ventricular block of any degree, serious arrhythmia or history of any one or more of the following cardiovascular conditions within the past 6 months: cardiac angioplasty or stenting, myocardial infarction, unstable angina, symptomatic peripheral vascular disease, coronary artery by-pass graft surgery, class II, III or IV congestive heart failure as defined by the New York Heart Association (NYHA)
* Active infection requiring antibiotics.
* History of cerebrovascular accident, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months
* History of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C.
* Patients who had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Subjects with < Grade 2 neuropathy or ≤ Grade 2 alopecia are an exception to this criterion and may qualify for the study.
* Patients with evidence of interstitial lung disease.
* Major surgical procedure, open biopsy, or significant traumatic injury within 3 weeks prior to beginning therapy, or anticipation of the need for a major surgical procedure during the course of the study; minor surgical procedures such as fine needle aspiration or core biopsy within 1 week prior to beginning therapy are also excluded.
* Known hypersensitivity to the study drugs or to drugs with similar chemical structures.
* Concurrent treatment with other experimental drugs.
* Participation in another clinical trial with any investigational drug within 30 days prior to study screening.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | from randomization to the date of radiological/clinical progression of disease or death, assessed up to 3 years
  The primary objective is to compare Decitabine plus Carboplatin combination versus physician' choice chemotherapy in terms of progression free survival

SECONDARY OUTCOMES:
Overall survival (OS) | from randomization to the date of death, assessed up to 3 years
  The secondary objective is to compare Decitabine plus Carboplatin combination versus physician' choice chemotherapy in terms of overall survival
Radiological response rate (in patients with measurable disease) | 3 years
  Radiological response rate
Duration of response | 3 years
  Duration of response
Cancer-Antigen 125 (CA-125) response rate per GCIG (Gynaecologic Cancer Intergroup) and change in CA-125 | 3 years
  Serum level of CA125 is used to monitor response to chemotherapy, relapse, and disease progression in ovarian cancer patients.
Toxicity profile | 3 years
  Incidence of adverse events
Patient Reported Outcome: Physical well-being | 3 years
  will be evaluated using the Functional Assessment of Cancer Therapy (FACT-O) and FACT-O Ovarian Cancer-specific Subscale (OCS) questionnaire. The total scores of both scales will be calculated, the scores of each question at each time point and their difference from baseline will be summarized for each treatment group. At a given visit, the change and/or percent change from baseline will be compared between the randomized treatment groups using an ANCOVA test using the treatment as a categorical factor and baseline measurement for the parameter as a continuous covariate.
  The time to an event in PRO (Patient Reported Outcome) of worsening of disease symptoms will be defined as the time from randomization to a 4-point reduction in the FACT-O questionnaire. Patients without a 4-point reduction will be censored on the date of their last PRO evaluation. Patients that do not have both a baseline measurement and at least one post-baseline measurement will not be included.
Patient Reported Outcome: Social/family well-being | 3 years
  will be evaluated using the Functional Assessment of Cancer Therapy (FACT-O) and FACT-O ovarian cancer-specific subscale (OCS) questionnaire. The total scores of both scales will be calculated, the scores of each question at each time point and their difference from baseline will be summarized for each treatment group. At a given visit, the change and/or percent change from baseline will be compared between the randomized treatment groups using an ANCOVA test using the treatment as a categorical factor and baseline measurement for the parameter as a continuous covariate.
  The time to an event in PRO of worsening of disease symptoms will be defined as the time from randomization to a 4-point reduction in the FACT-O questionnaire. Patients without a 4-point reduction will be censored on the date of their last PRO evaluation. Patients that do not have both a baseline measurement and at least one post-baseline measurement will not be included.
Patient Reported Outcome: Functional well being | 3 years
  will be evaluated using the Functional Assessment of Cancer Therapy (FACT-O) and FACT-O ovarian cancer-specific subscale (OCS) questionnaire. The total scores of both scales will be calculated, the scores of each question at each time point and their difference from baseline will be summarized for each treatment group. At a given visit, the change and/or percent change from baseline will be compared between the randomized treatment groups using an ANCOVA test using the treatment as a categorical factor and baseline measurement for the parameter as a continuous covariate.
  The time to an event in PRO of worsening of disease symptoms will be defined as the time from randomization to a 4-point reduction in the FACT-O questionnaire. Patients without a 4-point reduction will be censored on the date of their last PRO evaluation. Patients that do not have both a baseline measurement and at least one post-baseline measurement will not be included.
Patient Reported Outcome: Emotional well being | 3 years
  will be evaluated using the Functional Assessment of Cancer Therapy (FACT-O) and FACT-O ovarian cancer-specific subscale (OCS) questionnaire. The total scores of both scales will be calculated, the scores of each question at each time point and their difference from baseline will be summarized for each treatment group. At a given visit, the change and/or percent change from baseline will be compared between the randomized treatment groups using an ANCOVA test using the treatment as a categorical factor and baseline measurement for the parameter as a continuous covariate.
  The time to an event in PRO of worsening of disease symptoms will be defined as the time from randomization to a 4-point reduction in the FACT-O questionnaire. Patients without a 4-point reduction will be censored on the date of their last PRO evaluation. Patients that do not have both a baseline measurement and at least one post-baseline measurement will not be included.

CONTACTS AND LOCATIONS:
Overall Officials: Domenica Lorusso, MD, Principal Investigator — National Cancer Institute (NCI); Domenica Lorusso, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kantarjian H, Oki Y, Garcia-Manero G, Huang X, O'Brien S, Cortes J, Faderl S, Bueso-Ramos C, Ravandi F, Estrov Z, Ferrajoli A, Wierda W, Shan J, Davis J, Giles F, Saba HI, Issa JP. Results of a randomized study of 3 schedules of low-dose decitabine in higher-risk myelodysplastic syndrome and chronic myelomonocytic leukemia. Blood. 2007 Jan 1;109(1):52-7. doi: 10.1182/blood-2006-05-021162. Epub 2006 Aug 1. PMID 16882708
- [Background] Matei DE, Nephew KP. Epigenetic therapies for chemoresensitization of epithelial ovarian cancer. Gynecol Oncol. 2010 Feb;116(2):195-201. doi: 10.1016/j.ygyno.2009.09.043. Epub 2009 Oct 24. PMID 19854495
- [Result] Bukowski RM, Ozols RF, Markman M. The management of recurrent ovarian cancer. Semin Oncol. 2007 Apr;34(2 Suppl 2):S1-15. doi: 10.1053/j.seminoncol.2007.03.012. No abstract available. PMID 17512352
- [Result] Vaughan S, Coward JI, Bast RC Jr, Berchuck A, Berek JS, Brenton JD, Coukos G, Crum CC, Drapkin R, Etemadmoghadam D, Friedlander M, Gabra H, Kaye SB, Lord CJ, Lengyel E, Levine DA, McNeish IA, Menon U, Mills GB, Nephew KP, Oza AM, Sood AK, Stronach EA, Walczak H, Bowtell DD, Balkwill FR. Rethinking ovarian cancer: recommendations for improving outcomes. Nat Rev Cancer. 2011 Sep 23;11(10):719-25. doi: 10.1038/nrc3144. PMID 21941283
- [Result] Longley DB, Johnston PG. Molecular mechanisms of drug resistance. J Pathol. 2005 Jan;205(2):275-92. doi: 10.1002/path.1706. PMID 15641020
- [Result] Sharma S, Kelly TK, Jones PA. Epigenetics in cancer. Carcinogenesis. 2010 Jan;31(1):27-36. doi: 10.1093/carcin/bgp220. Epub 2009 Sep 13. PMID 19752007
- [Result] Das PM, Singal R. DNA methylation and cancer. J Clin Oncol. 2004 Nov 15;22(22):4632-42. doi: 10.1200/JCO.2004.07.151. PMID 15542813
- [Result] Ehrlich M. DNA hypomethylation in cancer cells. Epigenomics. 2009 Dec;1(2):239-59. doi: 10.2217/epi.09.33. PMID 20495664
- [Result] Taby R, Issa JP. Cancer epigenetics. CA Cancer J Clin. 2010 Nov-Dec;60(6):376-92. doi: 10.3322/caac.20085. Epub 2010 Oct 19. PMID 20959400
- [Result] Peedicayil J. The role of DNA methylation in the pathogenesis and treatment of cancer. Curr Clin Pharmacol. 2012 Nov;7(4):333-40. doi: 10.2174/157488412803305858. PMID 22794162
- [Result] Sang M, Wu X, Fan X, Sang M, Zhou X, Zhou N. Multiple MAGE-A genes as surveillance marker for the detection of circulating tumor cells in patients with ovarian cancer. Biomarkers. 2014 Feb;19(1):34-42. doi: 10.3109/1354750X.2013.865275. Epub 2013 Dec 10. PMID 24320162
- [Result] Gurion R, Vidal L, Gafter-Gvili A, Belnik Y, Yeshurun M, Raanani P, Shpilberg O. 5-azacitidine prolongs overall survival in patients with myelodysplastic syndrome--a systematic review and meta-analysis. Haematologica. 2010 Feb;95(2):303-10. doi: 10.3324/haematol.2009.010611. Epub 2009 Sep 22. PMID 19773261
- [Result] Balch C, Huang TH, Brown R, Nephew KP. The epigenetics of ovarian cancer drug resistance and resensitization. Am J Obstet Gynecol. 2004 Nov;191(5):1552-72. doi: 10.1016/j.ajog.2004.05.025. PMID 15547525
- [Result] Kelly TK, De Carvalho DD, Jones PA. Epigenetic modifications as therapeutic targets. Nat Biotechnol. 2010 Oct;28(10):1069-78. doi: 10.1038/nbt.1678. PMID 20944599
- [Result] Blum W, Klisovic RB, Hackanson B, Liu Z, Liu S, Devine H, Vukosavljevic T, Huynh L, Lozanski G, Kefauver C, Plass C, Devine SM, Heerema NA, Murgo A, Chan KK, Grever MR, Byrd JC, Marcucci G. Phase I study of decitabine alone or in combination with valproic acid in acute myeloid leukemia. J Clin Oncol. 2007 Sep 1;25(25):3884-91. doi: 10.1200/JCO.2006.09.4169. Epub 2007 Aug 6. PMID 17679729
- [Result] Wang LX, Mei ZY, Zhou JH, Yao YS, Li YH, Xu YH, Li JX, Gao XN, Zhou MH, Jiang MM, Gao L, Ding Y, Lu XC, Shi JL, Luo XF, Wang J, Wang LL, Qu C, Bai XF, Yu L. Low dose decitabine treatment induces CD80 expression in cancer cells and stimulates tumor specific cytotoxic T lymphocyte responses. PLoS One. 2013 May 9;8(5):e62924. doi: 10.1371/journal.pone.0062924. Print 2013. PMID 23671644
- [Result] Wijermans P, Lubbert M, Verhoef G, Bosly A, Ravoet C, Andre M, Ferrant A. Low-dose 5-aza-2'-deoxycytidine, a DNA hypomethylating agent, for the treatment of high-risk myelodysplastic syndrome: a multicenter phase II study in elderly patients. J Clin Oncol. 2000 Mar;18(5):956-62. doi: 10.1200/JCO.2000.18.5.956. PMID 10694544
- [Result] Plumb JA, Strathdee G, Sludden J, Kaye SB, Brown R. Reversal of drug resistance in human tumor xenografts by 2'-deoxy-5-azacytidine-induced demethylation of the hMLH1 gene promoter. Cancer Res. 2000 Nov 1;60(21):6039-44. PMID 11085525
- [Result] Watts GS, Futscher BW, Holtan N, Degeest K, Domann FE, Rose SL. DNA methylation changes in ovarian cancer are cumulative with disease progression and identify tumor stage. BMC Med Genomics. 2008 Sep 30;1:47. doi: 10.1186/1755-8794-1-47. PMID 18826610
- [Result] Barton CA, Hacker NF, Clark SJ, O'Brien PM. DNA methylation changes in ovarian cancer: implications for early diagnosis, prognosis and treatment. Gynecol Oncol. 2008 Apr;109(1):129-39. doi: 10.1016/j.ygyno.2007.12.017. Epub 2008 Jan 29. PMID 18234305
- [Result] Ibanez de Caceres I, Battagli C, Esteller M, Herman JG, Dulaimi E, Edelson MI, Bergman C, Ehya H, Eisenberg BL, Cairns P. Tumor cell-specific BRCA1 and RASSF1A hypermethylation in serum, plasma, and peritoneal fluid from ovarian cancer patients. Cancer Res. 2004 Sep 15;64(18):6476-81. doi: 10.1158/0008-5472.CAN-04-1529. PMID 15374957
- [Result] Li Y, Hu W, Shen DY, Kavanagh JJ, Fu S. Azacitidine enhances sensitivity of platinum-resistant ovarian cancer cells to carboplatin through induction of apoptosis. Am J Obstet Gynecol. 2009 Feb;200(2):177.e1-9. doi: 10.1016/j.ajog.2008.08.030. Epub 2008 Dec 25. PMID 19110234
- [Result] Frost P, Abbruzzese JL, Hunt B, Lee D, Ellis M. Synergistic cytotoxicity using 2'-deoxy-5-azacytidine and cisplatin or 4-hydroperoxycyclophosphamide with human tumor cells. Cancer Res. 1990 Aug 1;50(15):4572-7. PMID 1695122
- [Result] Jones PA, Baylin SB. The epigenomics of cancer. Cell. 2007 Feb 23;128(4):683-92. doi: 10.1016/j.cell.2007.01.029. PMID 17320506
- [Result] Stewart DJ. Mechanisms of resistance to cisplatin and carboplatin. Crit Rev Oncol Hematol. 2007 Jul;63(1):12-31. doi: 10.1016/j.critrevonc.2007.02.001. Epub 2007 Mar 1. PMID 17336087
- [Result] Gomyo Y, Sasaki J, Branch C, Roth JA, Mukhopadhyay T. 5-aza-2'-deoxycytidine upregulates caspase-9 expression cooperating with p53-induced apoptosis in human lung cancer cells. Oncogene. 2004 Sep 2;23(40):6779-87. doi: 10.1038/sj.onc.1207381. PMID 15273730
- [Result] Schwartsmann G, Schunemann H, Gorini CN, Filho AF, Garbino C, Sabini G, Muse I, DiLeone L, Mans DR. A phase I trial of cisplatin plus decitabine, a new DNA-hypomethylating agent, in patients with advanced solid tumors and a follow-up early phase II evaluation in patients with inoperable non-small cell lung cancer. Invest New Drugs. 2000 Feb;18(1):83-91. doi: 10.1023/a:1006388031954. PMID 10830142
- [Result] Pohlmann P, DiLeone LP, Cancella AI, Caldas AP, Dal Lago L, Campos O Jr, Monego E, Rivoire W, Schwartsmann G. Phase II trial of cisplatin plus decitabine, a new DNA hypomethylating agent, in patients with advanced squamous cell carcinoma of the cervix. Am J Clin Oncol. 2002 Oct;25(5):496-501. doi: 10.1097/00000421-200210000-00015. PMID 12393992
- [Result] Appleton K, Mackay HJ, Judson I, Plumb JA, McCormick C, Strathdee G, Lee C, Barrett S, Reade S, Jadayel D, Tang A, Bellenger K, Mackay L, Setanoians A, Schatzlein A, Twelves C, Kaye SB, Brown R. Phase I and pharmacodynamic trial of the DNA methyltransferase inhibitor decitabine and carboplatin in solid tumors. J Clin Oncol. 2007 Oct 10;25(29):4603-9. doi: 10.1200/JCO.2007.10.8688. PMID 17925555
- [Result] Fang F, Balch C, Schilder J, Breen T, Zhang S, Shen C, Li L, Kulesavage C, Snyder AJ, Nephew KP, Matei DE. A phase 1 and pharmacodynamic study of decitabine in combination with carboplatin in patients with recurrent, platinum-resistant, epithelial ovarian cancer. Cancer. 2010 Sep 1;116(17):4043-53. doi: 10.1002/cncr.25204. PMID 20564122
- [Result] Glasspool RM, Brown R, Gore ME, Rustin GJ, McNeish IA, Wilson RH, Pledge S, Paul J, Mackean M, Hall GD, Gabra H, Halford SE, Walker J, Appleton K, Ullah R, Kaye S; Scottish Gynaecological Trials Group. A randomised, phase II trial of the DNA-hypomethylating agent 5-aza-2'-deoxycytidine (decitabine) in combination with carboplatin vs carboplatin alone in patients with recurrent, partially platinum-sensitive ovarian cancer. Br J Cancer. 2014 Apr 15;110(8):1923-9. doi: 10.1038/bjc.2014.116. Epub 2014 Mar 18. PMID 24642620
- [Result] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Result] Pignata S, Lorusso D, Scambia G, Sambataro D, Tamberi S, Cinieri S, Mosconi AM, Orditura M, Brandes AA, Arcangeli V, Panici PB, Pisano C, Cecere SC, Di Napoli M, Raspagliesi F, Maltese G, Salutari V, Ricci C, Daniele G, Piccirillo MC, Di Maio M, Gallo C, Perrone F; MITO 11 investigators. Pazopanib plus weekly paclitaxel versus weekly paclitaxel alone for platinum-resistant or platinum-refractory advanced ovarian cancer (MITO 11): a randomised, open-label, phase 2 trial. Lancet Oncol. 2015 May;16(5):561-8. doi: 10.1016/S1470-2045(15)70115-4. Epub 2015 Apr 14. PMID 25882986